CLINICAL TRIAL: NCT01209065
Title: Phase I, Open Label, Two Period Study to Evaluate the Effects of Fosamprenavir/Ritonavir on GSK1349572 Pharmacokinetics and a Phase I, Randomized, Three-Way Crossover Study to Evaluate the Relative Bioavailability of Three Tablet Variants Made Using Micronized, Unmicronized and Intermediate Particle Sizes of GSK1349572 in Healthy Adult Subjects
Brief Title: GSK1349572 Drug Interaction Study With Fosamprenavir/Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113068
Record Dates: First submitted 2010-08-30; First posted 2010-09-24 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Infections, Human Immunodeficiency Virus and Herpesviridae
Keywords: integrase; fosamprenavir; ritonavir; GSK1349572
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; fosamprenavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Approximately 12 subjects will be enrolled. In the first treatment period, all subjects will receive GSK1349572 50 mg every 24 hours for 5 days. In Period 2, subjects will receive GSK1349572 50 mg every 24 hours in combination with fosamprenavir 700 mg plus ritonavir 100 mg every 12 hours for 10 days. Day 1 of Period 2 will be the day after Day 5 of Period 1. Subjects will have a screening visit within 30 days prior to the first dose of study drug, two treatment periods, and a follow-up visit 7-14 days after the last dose of study drug.
  Interventions: Drug: GSK1349572; Drug: Fosamprenavir; Drug: Ritonavir
- Part B (Experimental): Approximately 15 subjects will be enrolled and receive three single doses of GSK1349572 approximately one week apart. One will be the current tablet formulation containing micronized drug substance and 2 will be new tablet versions, one containing unmicronized drug substance and one containing an intermediate particle size drug substance. Subjects will have a screening visit within 30 days prior to the first dose of study drug, three treatment periods, and a follow-up visit 7-14 days after the last dose of study drug.
  Interventions: Drug: GSK1349572

INTERVENTIONS:
Drug: GSK1349572 — GSK1349572 is an integrase inhibitor being developed for the treatment of human immunodeficiency virus -1 infection by ViiV Healthcare. This drug is experimental and has not been approved by the Food and Drug Administration (FDA).
Drug: Fosamprenavir — Fosamprenavir is a drug in the protease inhibitor class that is approved by the FDA for the treatment of HIV infection.
  Other Names: TELZIR; LEXIVA; GW433908
  Arms: Part A
Drug: Ritonavir — Ritonavir is a drug in the protease inhibitor class that is approved by the FDA for the treatment of HIV infection.
  Other Names: NORVIR
  Arms: Part A

SUMMARY:
GSK1349572 is an integrase inhibitor being developed for the treatment of human immunodeficiency virus (HIV)-1 infection by GlaxoSmithKline (GSK) on behalf of Shionogi-ViiV HealthcareLLC. In HIV-infected patients where combination antiretroviral therapy is the standard of care, it is likely that it will be dosed with boosted protease inhibitors (PIs) including fosamprenavir/ritonavir (FPV/RTV or FPV/r). As FPV and RTV are modulators (induction as well as inhibition) of Uridine diphosphate glucuronosyltransferase (UGT) and Cytochrome P450 (CYP)3A which are the primary and secondary metabolic pathways of GKS1349572, it is likely that FPV/RTV will affect the pharmacokinetics (PK) of GSK1349572, therefore a drug interaction study is warranted and will be evaluated in Part A of this study. Part B will evaluate the effect of particle size of tablet variants on the PK of GSK1349572.

In Part A, approximately 12 subjects will receive GSK1349572 50mg every 24 hours (q24h) for 5 days (Treatment A). Subjects will then be administered GSK1349572 50mg q24h in combination with FPV/RTV 700/100 mg every 12 hours (q12h) (Treatment B) for 10 days. There will be no washout between treatments. In Part B 15 subjects will receive a single 50 mg dose (2 x 25mg tablet) in 3 different tablet variants of the same formulation, differing only in particle sizes of GSK1349572, under fasted conditions in a three-way crossover design. Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 7-14 days after the last dose of study drug.

DETAILED DESCRIPTION:
Official Study Title: Phase I, open label, two period, study to evaluate the effects of fosamprenavir/ritonavir on GSK1349572 pharmacokinetics and a phase I, randomized, three-way crossover study to evaluate the relative bioavailability of three tablet variants made using micronized, unmicronized and intermediate particle sizes of GSK1349572 in healthy adult subjects (ING113068).

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and bilirubin less than 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<146.8 pmol/L) is confirmatory]. or Child-bearing potential with a negative pregnancy test at both Screening and Day -1 and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Body weight greater than 50 kg for males and 45 kg for females and BMI within the range 18.5- 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug (including sulfa drugs) or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. History of sulphonamide allergy (FPV includes a sulphonamide moiety)
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, lower or upper gastrointestinal bleed, inflammatory bowel disease or pancreatitis should be excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of Gilbert's disease.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening electrocardiogram as listed in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Plasma GSK1349572 steady-state AUC(0-tau), Cmax, C0, Ctau, and Cmin following administration of GSK1349572 50 mg q24h for 5 days and following co-administration with FPV/RTV 700/100 mg q12h for 10 days | 15 days
Plasma GSK1349572 AUC(0-infinity), AUC(0-t), and Cmax following a single dose of GSK1349572 50 mg | 48 hours

SECONDARY OUTCOMES:
Safety and tolerability parameters, including adverse events, concurrent medication, clinical laboratory tests, ECG, and vital signs assessments | 15 days
Plasma amprenavir (APV) steady-state AUC(0-tau), Cmax, C0, Ctau, t½, and CL/F following administration of GSK1349572 50 mg q24h co-administered with FPV/RTV 700/100 mg q12h for 10 days | 15 days
Plasma GSK1349572 steady-state tmin, t1/2 and CL/F following administration of GSK1349572 50 mg q24h for 5 days and following co-administration with FPV/RTV 700/100 mg q12h for 10 days | 15 days
Plasma GSK1349572 C24, t1/2, tlag, tmax, CL/F and Vz/F following a single dose of GSK1349572 50 mg | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- [Derived] Song I, Borland J, Chen S, Peppercorn A, Wajima T, Piscitelli SC. Effect of fosamprenavir-ritonavir on the pharmacokinetics of dolutegravir in healthy subjects. Antimicrob Agents Chemother. 2014 Nov;58(11):6696-700. doi: 10.1128/AAC.03282-14. Epub 2014 Aug 25. PMID 25155604